CLINICAL TRIAL: NCT05497414
Title: Identifying Brain Dynamics Underlying Sleep and Mood in Depression
Brief Title: Neuroimaging Sleep and Mood in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Collaborators: One Mind (Unknown); Brain & Behavior Research Foundation (Other); 1907 Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 5562E
Record Dates: First submitted 2022-02-24; First posted 2022-08-11 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Two groups (healthy vs major depression) are studied under two conditions (rested vs sleep deprivation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep deprived (Experimental): Overnight sleep deprivation
  Interventions: Behavioral: Sleep deprivation
- Rested (No Intervention): Well-rested sleep pattern

INTERVENTIONS:
Behavioral: Sleep deprivation — Overnight sleep deprivation.
  Arms: Sleep deprived

SUMMARY:
This study will investigate how sleep and mood are related in patients with depression and in healthy controls. It will use MRI-based measures of brain function to determine how neural systems are modulated by sleep and sleep deprivation, and its links to mood in depression.

DETAILED DESCRIPTION:
The purpose of this work is to identify brain networks that underlie sleep and mood using a combination of EEG and fMRI. Sleep deprivation can elicit rapid improvements in mood in some patients with depression, while some patients do not show any significant changes in mood. We will image the brain while measuring physiological and electrical signals in healthy individuals and in patients with depression. Subjects will participate in combined EEG-MRI studies that will involve the use of perceptual and attentional tasks, and will involve recording physiological variables such as breathing, heart rate, eye movements, and blood pressure. If combined EEG-MRI cannot be completed due to data quality reasons, subjects will participate in EEG or MRI alone. Subjects will participate in a blood draw to assess for inflammatory markers related to mood. Subjects will be either well-rested or sleep deprived. For sleep deprivation, subjects will be asked to stay awake overnight under the supervision of a member of the study team at Boston University, and then would be asked to do an fMRI, EEG, or EEG-MRI scan. fMRI studies will be performed at the Boston University Center for Cognitive Neuroimaging. During the study visit, subjects will answer questions in structured interviews, will fill out questionnaires that will contain questions related to their mental health. Subjects will be shown visual stimuli and/or listen to auditory stimuli, and/or asked to perform simple behavioral tasks related to these stimuli. Some of the visual stimuli will be emotionally salient. Wrist actigraphy will be used to monitor sleep behavior. Remote daily mood and sleep assessments will be performed for up to two weeks prior to imaging. These assessments will be sent as emails or text messages to participants.

ELIGIBILITY:
Inclusion criteria:

* Adult aged 18-80

Inclusion criteria for patient cohort only:

- Current diagnosis of major depressive disorder

Exclusion criteria:

* Must not have ferrous metal implanted in head or body
* Must have no history of major head trauma
* Must not have implanted electronic devices (e.g., pacemaker, neurostimulator)
* Must not be pregnant, suspect they are pregnant, or seeking to become pregnant
* Must not be claustrophobic
* Must have no piercings or jewelry that cannot be removed
* Weight less than 250 pounds
* No lifetime history of schizophrenia or any other psychosis disorder, substantial intellectual disability, bipolar disorder, post-traumatic stress disorder or obsessive compulsive disorder
* No alcohol or substance abuse or dependence within the past 6 months
* No significant personality dysfunction
* Must not indicate significant suicide risk.
* Must not be taking medications that significantly affect sleep, psychiatric function, blood/vascular function, or anti-inflammatory medications (other than minor NSAID use).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in fMRI signals in thalamus region of interest (ROI) from baseline to post intervention | Through study completion (approximately 1 month)
  fMRI signal (units: %)
Change in fMRI signals in amygdala ROI from baseline to post intervention | Through study completion (approximately 1 month)
  fMRI signal (units: %)
Change in tasked evoked responses in amygdala ROI from baseline to post intervention | Through study completion (approximately 1 month)
  Task evoked responses in amygdala ROI (units: %)
Change in cerebrospinal fluid (CSF) flow measurements from baseline to post intervention | Through study completion (approximately 1 month)
  Fluid flow measured with MRI (units: %)
Change in Montgomery-Asberg Depression Rating from baseline to post intervention | Through study completion (approximately 1 month)
  Mood scores, measured on scale of 0-60
Change in whole-brain voxelwise fMRI activity from baseline to post intervention | Through study completion (approximately 1 month)
  fMRI measure of hemodynamics (units: %)

SECONDARY OUTCOMES:
Change in EEG dynamics from baseline to post intervention | Through study completion (approximately 1 month)
  Amplitude of EEG signals (units: uV^2)
Change in dot probe task performance from baseline to post intervention | Through study completion (approximately 1 month)
  Behavior on emotional task (units: ms)
Change in blood biomarkers of C-reactive protein from baseline to post intervention | Through study completion (approximately 1 month)
  Blood analysis results (units: mg/L)
Change in blood levels of Interleukin 6 from baseline to post intervention | Through study completion (approximately 1 month)
  Measured in pg/mL
Change in Magnetic Resonance Spectroscopy (MRS) measurement of lactate from baseline to post intervention | Through study completion (approximately 1 month)
  MRS measure of lactate (units: i.u.)
Change in MRS measurement of myo-inositol from baseline to post intervention | Through study completion (approximately 1 month)
  Magnetic Resonance Spectroscopy measure of myo-inositol (units: i.u.)
Change in Positive and Negative Affect Scale 21 (PANAS-21) rating from baseline to post intervention | Through study completion (approximately 1 month)
  The Positive and Negative Affect Scale (PANAS-21) assess positive and negative affect using scales relating to how participants feel about certain words.
Change in Positive and Negative Affect Scale 21 (PANAS-21) rating during intervention | Throughout intervention (approximately 17 hours)
  The Positive and Negative Affect Scale (PANAS-21) assess positive and negative affect using scales relating to how participants feel about certain words.
Change in Shame Inventory rating from baseline to post intervention | Through study completion (approximately 1 month)
  The Shame Inventory assess participants' feelings related to shame. Units: scale.
Change in Shame Inventory rating during intervention | Throughout intervention (approximately 17 hours)
  The Shame Inventory assess participants' feelings related to shame. Units: scale.
Change in Anxiety Sensitivity Index (ASI-3) rating from baseline to post intervention | Through study completion (approximately 1 month)
  The Anxiety Sensitivity Index assess participants' concern related to anxiety.Units: scale.
Change in Anxiety Sensitivity Index (ASI-3) rating during intervention | Throughout intervention (approximately 17 hours)
  The Anxiety Sensitivity Index assess participants' concern related to anxiety.Units: scale.
Change in Depression, Anxiety, and Stress Scale (DASS-21) rating from baseline to post intervention | Through study completion (approximately 1 month)
  The Depression, Anxiety, and Stress Scale assesses participants emotional states. Units: scale.
Change in Depression, Anxiety, and Stress Scale (DASS-21) rating during intervention | Throughout intervention (approximately 17 hours)
  The Depression, Anxiety, and Stress Scale assesses participants emotional states. Units: scale.
Patient health questionnaire (PHQ-9) | Pre-enrollment
  This patient health questionnaire is used to compute a general depression score.Units: scale.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lewis, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States